CLINICAL TRIAL: NCT04758598
Title: The Effects of DSLT and SLT on the Corneal Endothelium: A GLAUrious Trial Sub-Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BelkinVision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2020-01
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2021-02

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: DSLT treatment vs. SLT treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Selective Laser Trabeculoplasty (DSLT) (Experimental): Direct Selective Laser Trabeculoplasty (DSLT): employs frequency-doubled, Q-switched Nd:YAG laser with a wavelength of 532 nm. During the procedure, a laser beam targets the trabecular meshwork (TM) - to improve intraocular fluid outflow. The laser beam is delivered in short nanosecond pulses and the selective cellular effect occurs at the pigmented cells of the TM. This increases the permeability of the TM endothelial cells and thereby increases outflow, resulting in reductions in IOP. In contrast to SLT, the DSLT treatment directs the laser beam directly through the sclera around the limbus without the need for a delivery device (gonioscope lens). Laser treatment lasts for about 2 seconds with about 120 laser shots delivered to the sclera around the limbus.
  Interventions: Device: Direct Selective Laser Trabeculoplasty (DSLT)
- Selective Laser Trabeculoplasty (SLT) (Active Comparator): SLT employs frequency doubled Q switched Nd:YAG laser with a wavelength of 532 nm. It is delivered in short nano second pulses and the resulting selective effect to the pigmented cells of the TM, leaving the surrounding non-pigmented cells unaffected. This increases the permeability of the TM endothelial cells and can assist in increasing outflow and hence result in reductions in IOP. The procedure lasts approximately 10 minutes, with delivering 100 separate laser beams through a manually rotated mirrored lens (gonioscope), involving prolonged contact with the participant's eye. This treatment is applied on the cornea through a gonioscopic lens which is used to direct the laser beam to the desired location - the TM (360 degrees of treatment area).
  Interventions: Device: Selective Laser Trabeculoplasty (SLT)

INTERVENTIONS:
Device: Direct Selective Laser Trabeculoplasty (DSLT) — DSLT employs frequency-doubled, Q-switched Nd:YAG laser with a wavelength of 532 nm. During the procedure, a laser beam targets the trabecular meshwork (TM) - to improve intraocular fluid outflow. The laser beam is delivered in short nanosecond pulses and the selective cellular effect occurs at the pigmented cells of the TM. This increases the permeability of the TM endothelial cells and thereby increases outflow, resulting in reductions in IOP. In contrast to SLT, the DSLT treatment directs the laser beam directly through the sclera around the limbus without the need for a delivery device (gonioscope lens). Laser treatment lasts for about 2 seconds with about 120 laser shots delivered to the sclera around the limbus.
  Arms: Direct Selective Laser Trabeculoplasty (DSLT)
Device: Selective Laser Trabeculoplasty (SLT) — SLT employs frequency doubled Q switched Nd:YAG laser with a wavelength of 532 nm. It is delivered in short nano second pulses and the resulting selective effect to the pigmented cells of the TM, leaving the surrounding non-pigmented cells unaffected. This increases the permeability of the TM endothelial cells and can assist in increasing outflow and hence result in reductions in IOP. The procedure lasts approximately 10 minutes, with delivering 100 separate laser beams through a manually rotated mirrored lens (gonioscope), involving prolonged contact with the participant's eye. This treatment is applied on the cornea through a gonioscopic lens which is used to direct the laser beam to the desired location - the TM (360 degrees of treatment area).
  Arms: Selective Laser Trabeculoplasty (SLT)

SUMMARY:
The objective of this study is to compare the long-term (6 months) effects of Direct Selective Laser Trabeculoplasty (DSLT) treatment and SLT (Selective Laser Trabeculoplasty) treatment on corneal endothelial cell counts and corneal thickness.

DETAILED DESCRIPTION:
Rational:

SLT has known transient effect on corneal endothelial cell (CEC) counts yet no data is yet available with DSLT.

This study is relevant as the DSLT treatment area is at the limbus: CEC progenitor site

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years or older, with visual acuity > 6/60 in both eyes
2. Open angle glaucoma including exfoliative or pigmentary glaucoma or ocular hypertension.
3. IOP ≥ 22mmHg or ≤35mmHg (after washout of any IOP-lowering medications) for participants with open angle glaucoma or IOP ≥ 24mmHg to ≤35mmHg (after washout of any IOP-lowering medications) for participants with ocular hypertension
4. Gonioscopically visible scleral spur for 360 degrees without indentation
5. Ability to visualize the peri-limbal sclera for 360 degrees (using a speculum)
6. Willing and able to participate in the 12-month study, to comply with the study procedures and to adhere to the follow-up schedule.
7. Participant capable of giving informed consent

Exclusion Criteria:

1. Contraindications to conventional laser trabeculoplasty (e.g. corneal abnormalities etc.)
2. Angle Closure Glaucoma
3. Congenital or developmental glaucoma
4. Secondary glaucoma except exfoliative or pigmentary glaucoma
5. Inability to conduct a reliable visual field (defined as fixation losses, false positives or false negatives greater than 33%)
6. Presence of any Peripheral Anterior Synechiae (PAS) in the study eye
7. Any of the following visual field findings using the Humphrey visual field analyzer the SITA-standard 24-2 program:

   1. A visual field MD of worse than -12dB
   2. Greater than or equal to 75% of points depressed below the 5% level and greater than or equal to 50% of points depressed below the 1% level on the PD plot
   3. At least 50% of points (i.e., 2 or more) within the central 5 degrees with a sensitivity ≤0dB on the decibel plot
   4. Points within the central 5 degrees of fixation with a sensitivity <15 dB in both hemifields on the decibel plot
8. A visual field MD of worse than -12dB in the fellow eye
9. Cup:Disc Ratio more than 0.8
10. More than three hypotensive medications required (combination drops are considered 2 medications)
11. Prior incisional or laser glaucoma surgery (including previous SLT) in the study eye
12. Prior corneal refractive surgery
13. Complicated cataract surgery ≤ 6 months prior to enrollment
14. Presence of visually significant cataract in the opinion of the investigator
15. Clinically significant disease in either eye as determined by the Investigator
16. Clinically significant amblyopia in either eye
17. Dense pigmentation or haemorrhage in the peri-limbal conjunctiva or anterior sclera
18. Women who are pregnant or may become pregnant during the course of the study
19. In the opinion of the investigator the participant might require other ocular surgery within the 12-month follow-up period, unless for further reduction of their IOP.
20. Concurrent treatment with topical, nasal, inhaled or systemic steroids.
21. Uncontrolled systemic disease that could impact the ability of the participant to attend follow up visits as per the discretion of the investigator
22. Participation in another clinical study, not including a GLAUrious sub-study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Difference between the mean baseline and 6 month central corneal thickness, DSLT vs SLT | 6 months
  Central corneal thickness will be assessed by pachymetry
Difference between the mean baseline and 6 month corneal endothelial cell count, DSLT vs SLT | 6 months
  Corneal endothelial cell count will be assessed with specular microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Akhali Mzera Eye Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share the protocol, statistical plan and results